CLINICAL TRIAL: NCT03477630
Title: Open Treatment for Pain and Inflammation in Knee Osteoarthrosis With Platelet-rich Plasma, Comparative Study With Hyaluronic Acid
Brief Title: Treatment of Osteoarthrosis of the Knee With Platelet Rich Plasma, Comparative Study With Hyaluronic Acid
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Karla Andrea Arias Varela (Individual)
Responsible Party: Sponsor-Investigator, Karla Andrea Arias Varela, Clinical Research, Varela, Karla Andrea Arias, M.D.
Organization: Varela, Karla Andrea Arias, M.D. (Individual)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: PRP 3.5 - 01 version 1.3
Record Dates: First submitted 2018-03-12; First posted 2018-03-26 (Actual); Last update posted 2022-06-16 (Actual); Status verified 2022-06

CONDITIONS: Osteoarthritis
Keywords: gonarthrosis
MeSH Terms: conditions — Osteoarthritis; Osteoarthritis, Knee | interventions — Hyaluronic Acid

STUDY DESIGN:
Intervention Model Description: Open, cohort, prospective controlled, randomized study with one year of follow-up.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Platelet Rich Plasma (Experimental): Four intra-articular infiltration of autologous PRP every 15 days.
  Interventions: Biological: Platelet Rich Plasma
- Hyaluronic Acid (Active Comparator): One intra-articular infiltration of SYNVISC-ONE
  Interventions: Drug: Hyaluronic Acid

INTERVENTIONS:
Biological: Platelet Rich Plasma — intra-articular infiltration of 8 ml of autologous PRP every 15 days.
  Other Names: PRP
  Arms: Platelet Rich Plasma
Drug: Hyaluronic Acid — intra-articular infiltration of a single dose of HA
  Other Names: HA
  Arms: Hyaluronic Acid

SUMMARY:
To compare changes in functionality and pain level using questionnaires EVA, Lequesne and WOMAC in patients treated with 4 doses of 8 ml of autologous Platelet Rich Plasma every 15 days applied through intra-articular infiltration and patients treated with an intra-articular infiltration of 1 dose of SYNVISC-ONE ® 6 ml pre-filled syringe, placed according to standard protocol, in patients with OA grade II-IV.

DETAILED DESCRIPTION:
28 participants with grade II-IV knee OA who met all the inclusion criteria and none of the exclusion criteria were recruited and selected. They were randomized into two groups, one received 4 doses of PRP and the other conventional hyalurinic acid treatment. Each patient underwent an evaluation of their baseline condition and physical examination of the affected knee by applying the functional and pain level questionnaires: WOMAC, VAS and LEQUESNE, after which each of the treatments was applied, respectively. The control group received 1 dose of SYNVISC-ONE, placed according to the standard intra-articular infiltration protocol, and group 2 received 4 intra-articular infiltrations of activated autologous PRP placed every 15 days. The patients were assessed at 3, 6 and 12 months by physical examination and the same surveys were applied to determine the progress and efficacy of the treatments using the same surveys. Finally, a statistical analysis was performed to compare the results between the two treatments.

ELIGIBILITY:
Inclusion Criteria

1. Osteoarthrosis grade II, III and IV of Kellgren and Lawrence
2. Chronic painful knee of mechanical characteristics.
3. Absence of local or systemic septic process.
4. Hematological and biochemical blood analysis without alterations that contraindicate the treatment.
5. Informed consent in writing from the patient.
6. Patient able to understand the nature of the study

Exclusion Criteria:

1. Allergic to egg
2. Alteration in blood tests for platelets count in whole blood (hemogram)
3. Patients presenting positive serology for HIV 1 and 2, Hepatitis B [HBsAg, Anti-HBV-Ab], Hepatitis C [Anti-HCV-Ab] and VDRL ).
4. Participant who presents platelets in the peripheral blood outside the range of normality (150.00 to 450,000).
5. Patients with positive serology for HIV 1, and 2, VDRL, Hepatitis B [HBsAg, Anti HBs] Hepatitis C (HCV).
6. Simultaneous participation in another clinical trial or treatment with another product in the experimental phase in the 30 days prior to inclusion in the study.
7. Neoplastic disease
8. Immunosuppressive states.
9. Other pathologies or circumstances that compromise participation in the study according to medical criteria.
10. The participant who has received intra-articular injection in knee with steroid deposit in the last 3 months. .
11. Participant with religious or cultural conflicts due to the use of Platelet Rich Plasma.
12. Participant with an activev infectious diseases in blood.
13. Patients with anticoagulant treatment (warfarin, heparin) in the last 6 months.
14. Participant with a history of skin, muscle or bone cancer in the lower limbs.
15. Participant with psychological, emotional, social problems or any other situation that may interfere with the requirements of the study.
16. Participant hospitalized for medical or surgical reasons.
17. Participants with an arthroscopy in the last 6 months.
18. Participants with severe osteoarthritis of the knee (Varo or Valgo)

Ages: 40 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2019-02-14 (Actual); Primary Completion 2020-07-25 (Actual); Study Completion 2020-09-16 (Actual)

PRIMARY OUTCOMES:
Changes in pain levels and functionality | Baseline, 3 months, 6 months and 12 months.
  Eva scale for the intensity of pain associated with activities of daily living and if sports activities are practiced. Lequesne index for knee osteoarthritis and physical function, pain and stiffness measured by Womac index.Each of the 3 questionnaires was evaluated at four different times: baseline, 3 months, 6 months and 12 months after treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Carlos Palavicini, Study Director — FIFA MD
Locations (1):
- Hospital Clínica Bíblica, San José, Costa Rica

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Riboh JC, Saltzman BM, Yanke AB, Fortier L, Cole BJ. Effect of Leukocyte Concentration on the Efficacy of Platelet-Rich Plasma in the Treatment of Knee Osteoarthritis. Am J Sports Med. 2016 Mar;44(3):792-800. doi: 10.1177/0363546515580787. Epub 2015 Apr 29. PMID 25925602
- [Background] Carrillo-Mora P, Gonzalez-Villalva A, Macias-Hernandez SI, Villasenor CP. [Platelets-rich plasma: a versatile tool for regenerative medicine?]. Cir Cir. 2013 Jan-Feb;81(1):74-82. Spanish. PMID 23461926
- [Background] Shahid M, Kundra R. Platelet-rich plasma (PRP) for knee disorders. EFORT Open Rev. 2017 Mar 13;2(1):28-34. doi: 10.1302/2058-5241.2.160004. eCollection 2017 Jan. PMID 28607768
- [Result] Raeissadat SA, Rayegani SM, Hassanabadi H, Fathi M, Ghorbani E, Babaee M, Azma K. Knee Osteoarthritis Injection Choices: Platelet- Rich Plasma (PRP) Versus Hyaluronic Acid (A one-year randomized clinical trial). Clin Med Insights Arthritis Musculoskelet Disord. 2015 Jan 7;8:1-8. doi: 10.4137/CMAMD.S17894. eCollection 2015. PMID 25624776